CLINICAL TRIAL: NCT04691336
Title: Piloto Study of an Individualized Plan for Improving Adherence to Portable Oxygen Therapy in Patients With Respiratory Pathology
Brief Title: Individualized Plan for Improving Adherence to Portable Oxygen Therapy in Patients With Respiratory Pathology
Acronym: PIMAOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Liquide Healthcare Spain (Industry)
Collaborators: Hospital Sant Joan de Deu (Other)
Responsible Party: Principal Investigator, David Rudilla, Principal investigator, Air Liquide Healthcare Spain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIMAOX-CEI 20/04
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: COPD; ILD; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PIMAGroup (Experimental): All patients were summoned to the care center, being evaluated individually by a nurse, and based on the results, a care plan adapted to the specific needs and objectives was initiated. This care plan involved monitoring using different channels (face-to-face, telephone), with the main objective of monitoring the evolution of compliance, adherence and improving the quality of life of patients. The interventions that were carried out were educational and formative (using counseling communication skills), and technological (using monitoring tools in specific cases). The empowerment program was an educational session in which the nurse discussed content about dyspnea, the benefits of therapy, etc.
  Interventions: Behavioral: Educational and Training with counselling

INTERVENTIONS:
Behavioral: Educational and Training with counselling — The nurse conducts a structured interview that covers the following areas: information on respiratory attraction and the symptom of dyspnea, expectations and beliefs about oxygen therapy, use of oxygen therapy, healthy habits, social support. It also evaluates the patient's perception of oxygen therapy, and the level of dyspnea using the mMRC scale. After this, the nurse evaluates the current level of adherence, and if she considers that the patient needs a reinforcement session, she schedules a workshop with 3 other patients and their main caregivers. This workshop takes place 30 days after this interview. In other patients, depending on the level of adherence, a support call is made, and all patients are visited again at the center at 90 days, performing the same evaluation with a structured interview and the scales that were made on day 1

SUMMARY:
Pilot study with patients with prescription of portable oxygen therapy, to test the impact on adherence of a patient-centered empowerment program, with contents on the nature of the respiratory pathology, the symptom of dyspnea, the benefits of the therapy, adjustment expectations and beliefs, as well as health habits.

DETAILED DESCRIPTION:
All patients were summoned to the care center, being evaluated individually by a nurse, and based on the results, a care plan adapted to the specific needs and objectives was initiated. This care plan involved monitoring using different channels (face-to-face, telephone), with the main objective of monitoring the evolution of compliance, adherence and improving the quality of life of patients. The interventions that were carried out were educational and formative (using counseling communication skills), and technological (using monitoring tools in specific cases). The empowerment program was an educational session in which the nurse discussed content about dyspnea, the benefits of therapy, etc.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years old) with prescription of portable oxygen therapy by the Pneumology Service of the Sant Joan de Dèu Hospital in Manresa.

Exclusion Criteria:

* Psychophysical inability to carry out questionnaires or refusal to answer them.
* Severe displacement problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Adherence - Changes | Day 1 and Day 90
  Number of hours of use of oxygen concentrator / day
Dyspnea - Changes | Day 1 and Day 90
  Level of dyspnea, measured with the mMRC scale. Minimum score: 0, Maximum score: 4. A high score implies a worse outcome.
Quality of Life - Changes | Day 1 and Day 90
  General well-being state, measured with a visual analog scale. Minimum score: 0, Maximum score: 10. A high score implies a better outcome.
Emotional State - Changes | Day 1 and Day 90
  Mood, measured with a 3 level likert item . Minimum score: 0, Maximum score: 2. A high score implies a better outcome.
Activities | Day 1 and Day 90
  Level of activity. measured with a 3 level likert item . Minimum score: 0, Maximum score: 2. A high score implies a better outcome.
Social Relations | Day 1 and Day 90
  Level of social activity. measured with a 3 level likert item . Minimum score: 0, Maximum score: 2. A high score implies a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: David Rudilla, PhD, Principal Investigator — Air Liquide Healthcare
Locations (1):
- David Rudilla, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
1. Clinical impact, assistance and / or technological development. This project has a great impact and clinical and technological significance. From the clinical point of view, the aim is to identify the patient in order to better serve him and ensure adherence to one of the treatments where it is more complex to achieve patient compliance.
  2. Bibliometric impact. This project is expected to lead to world-class, high-impact publications.
Time Frame: 36 months after the publication of the work in a research journal
Access Criteria: Researchers who want to replicate the study

REFERENCES:
- [Background] Rudilla D, Valenzuela C, Beceiro MJ, Alonso T, Ancochea J. Fibrosis pulmonar idiopática y emociones. Una revisión sobre los aspectos psicológicos de la enfermedad. Rev Patol Respir. 2018; 21(2): 54-60
- [Background] Rudilla D, Oliver A, Galiana L, Barreto P. A new measure of home care patients' dignity at the end of life: The Palliative Patients' Dignity Scale (PPDS). Palliat Support Care. 2016 Apr;14(2):99-108. doi: 10.1017/S1478951515000747. Epub 2015 Jun 11. PMID 26062752